CLINICAL TRIAL: NCT06634186
Title: The Impact of a Dietary Fiber Enriched Diet on Frailty, Sarcopenia, Systemic Inflammation and Microbiome Composition in Patients with Liver Cirrhosis
Brief Title: The Impact of a Dietary Fiber Enriched Diet on the Outcome of Patients with Liver Cirrhosis
Acronym: ChainCirr
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 10928_BO_S_2023
Record Dates: First submitted 2024-07-18; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dietary intervention (Experimental): The studied patients will receive a dietary intervention. This intervention includes a dietary counselling, that enables our patients to establish a fiber-enriched diet. This adapted diet will be supplemented by the short-chain-fatty-acid propionate, that functions as fiber-surrogate.
  Interventions: Dietary Supplement: Dietary intervention

INTERVENTIONS:
Dietary Supplement: Dietary intervention — The aim of the dietary intervention is the implementation of a fiber-enriched diet. Therefore, patients receive dietary counseling, supplemented with propionate, that functions as fiber-surrogate.

SUMMARY:
The goal of this dietary intervention is to study the impact of a dietary fiber enriched diet on the intestinal dysbiosis, systemic inflammation and cirrhosis-related complications in patients with liver cirrhosis.

Therefore, our aim is to investigate the impact of a dietary fiber enriched diet on

* frailty and sarcopenia
* systemic inflammation
* microbiome composition
* quality of life and the composition of patients diet.

Participants receive a dietary counselling and will be asked to increase their dietary fiber intake. As malnutrition is a common complication in cirrhosis and patients with advanced liver disease often show a disability to meet their daily food-requirements, the recommended intake of 30 gram dietary fibers per day is unlikely in this group of patients. Therefore, the fiber-enriched diet will be supplemented by the physiological short-chain-fatty-acid propionate, as a fiber-surrogate.

DETAILED DESCRIPTION:
The disease course of liver cirrhosis is associated with a progressing dysbiosis of the intestinal microbiome and systemic inflammation, that leads to the development of cirrhosis-associated immune dysfunction (CAID). In healthy individuals, the microbiome uses orally incorporated dietary fibers for the production of short-chain-fatty-acids (SCFA). One of these physiological short-chain-fatty acids is propionate. SCFA´s are essential for a maintained integrity of the intestinal barrier and promote anti-inflammatory effects. Due to a reduction of symbiotic gut bacteria and an elevated number of potentially pathogenic microbes in cirrhosis, diminished levels of SCFA can be observed in this group of patients. Consequently, the permeability of the gut barrier increases and a bacterial translocation results. This translocation is a main driver of systemic inflammation and is linked to a higher likelihood for infections, such as spontaneous bacterial peritonitis (SBP). Furthermore, systemic inflammation promotes the degradation of skeleton muscles (sarcopenia) and frailty. Both are associated with a poor prognosis in cirrhosis. However, the impact of an adapted diet, that intends to normalize the intestinal SCFA-levels, on the clinical outcome of patients with advanced liver disease, needs to be further evaluated.

Therefore, the included patients receive dietary counseling, supplemented with propionate, that functions as fiber-surrogate. The dietary-intervention will last for a period of two months.

ELIGIBILITY:
Inclusion Criteria:

* Patients of legal age and with the ability to give informed consent
* Patients with liver cirrhosis and portal hypertension

Exclusion Criteria:

* Patients with transjugular intrahepatic portosystemic shunt (TIPS)
* significant immunosuppression
* malignant tumor
* underage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change of the Liver Frailty Index | The Liver Frailty Index will be measured at each study visit (Baseline, after 2 month and after 5 month)

SECONDARY OUTCOMES:
Change of phase angle (°) | Phase angle will be measured at each study visit (Baseline, after 2 month and after 5 month)
  The phase angle will be measured with body impedance analysis (BIA).
Change of systemic inflammation | Interleukin-6 will be measured at each study visit (Baseline, after 2 month and after 5 month)
  Measurement of interleukin-6
Change of microbiome composition | Stool samples will be collected at each study visit (Baseline, after 2 month and after 5 month)
Change of diet composition | Questionnaires will be collected at each study visit (Baseline, after 2 month and after 5 month)
  assessed with food-frequency-questionnaire (FFQ)
Change of body cell mass (BCM; kg) | BCM will be measured at each study visit (Baseline, after 2 month and after 5 month)
  Body cell mass will be measured with body impedance analysis (BIA)
Improvement of quality of life | Each study visit (Baseline, after 2 month and after 5 month)
  assessed with SF-36 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Hannover Medical School (MHH), Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided